CLINICAL TRIAL: NCT03884595
Title: Early Identification of Sepsis in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Michal Fedora, Assoc. prof. Michal Fedora, MD., Ph.D., Brno University Hospital
Other Study IDs: FNBRNO-2017/01
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Sepsis; Shock, Septic; Sepsis, Severe; SIRS
Keywords: sepsis; septic shock; severe sepsis; SIRS; children; immature platelet fraction (IPF); immature granulocytes (IG); nucleated red blood cells (NRBC)
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- No SIRS: Children without clinical signs of SIRS, according to Goldstein criteria.
  Interventions: Diagnostic Test: IG, IPF, NRBC, CRP, PCT, presepsin
- SIRS: Children with clinical signs of SIRS, according to Goldstein criteria.
  Interventions: Diagnostic Test: IG, IPF, NRBC, CRP, PCT, presepsin
- Sepsis: Children with clinical signs of sepsis, according to Goldstein criteria.
  Interventions: Diagnostic Test: IG, IPF, NRBC, CRP, PCT, presepsin
- Severe sepsis: Children with clinical signs of severe sepsis, according to Goldstein criteria.
  Interventions: Diagnostic Test: IG, IPF, NRBC, CRP, PCT, presepsin
- Septic Shock: Children with clinical signs of septic shock, according to Goldstein criteria.
  Interventions: Diagnostic Test: IG, IPF, NRBC, CRP, PCT, presepsin

INTERVENTIONS:
Diagnostic Test: IG, IPF, NRBC, CRP, PCT, presepsin — Assessment of blood cell count parameters and inflammation markers - IG, IPF, NRBC, CRP, PCT, presepsin according to study group.

SUMMARY:
This observational nation-wide study is focused on evaluation of the new possible biomarkers for pediatric sepsis and their specificity/sensitivity in combination with usual diagnostic markers for sepsis in the terms of early identification of sepsis, severe sepsis, and septic shock.

DETAILED DESCRIPTION:
The understanding of sepsis pathophysiology underwent a great progress during the last decades and the therapy of sepsis is in the focus of the research for many years, but sepsis is still one of the main causes of death in the ICUs around the world. Systemic inflammatory response syndrome (SIRS) is closely connected with the sepsis development, but SIRS also represents a high risk of organ dysfunction in non-infectious patients (trauma, stress, cardiopulmonary arrest). Early diagnosis and prevention of the organ dysfunction are the mainstay of the correct and timely therapy, but currently there is no reliable, quick and simple method for the diagnosis of sepsis. And also there is no generally accepted clinical or laboratory parameter, which can be used to differentiate between sepsis and SIRS.

There are some commonly available biomarkers that showed promising results in critically ill adult patients. Those include immature platelet fraction (IPF), immature granulocytes (IG) count and nucleated red blood cells (NRBC) count. The knowledge of their variability in different phases of illness (SIRS/sepsis/severe sepsis/septic shock) in pediatric patients is very limited, as is their connection with other generally used markers of infection (CRP, procalcitonin, presepsin).

This study is strictly non-interventional and focused on usability of above mentioned biomarkers in the early diagnosis of sepsis/SIRS and on the reduction of morbidity/mortality of pediatric intensive care unit (PICU) patients with sepsis/SIRS.

In all patients admitted to PICU in selected study period, the inflammation markers - C-reactive protein (CRP), procalcitonin (PCT), presepsin (soluble cluster of differentiation 14-subtypes) and full blood count parameters -IPF,IG,NRBC will be measured at the time of admission and on 3rd, 5th and 7th day of stay in intensive care. The organ dysfunction score will be evaluated daily.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to PICU until the 18th year of age
* expected length of stay > 48 hours

Exclusion Criteria:

* oncology patients
* immunosuppressive therapy
* immunostimulant therapy
* autoimmune disease
* post-organ transplant patient
* thrombocytopaenia, thrombocytopathy

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to PICU.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
IG and IPF concentration for early sepsis identification | 7 days
  The levels of IG and IPF will be obtained in first 7 days after admission. The IG and IPF will be evaluated for the possibility of early sepsis recognition.

SECONDARY OUTCOMES:
IG serum levels in patients with SIRS and sepsis/severe sepsis/septic shock | 7 days
  The levels of IG will be obtained in first 7 days after admission. The IG will be evaluated for the possibility of distinguish patients with or without SIRS and sepsis/severe sepsis/septic shock sepsis/septic shock.
IPF serum levels in patients with SIRS and sepsis/severe sepsis/septic shock | 7 days
  The levels of IPF will be obtained in first 7 days after admission. The IPF will be evaluated for the possibility of distinguish patients with or without SIRS and sepsis/severe sepsis/septic shock sepsis/septic shock.
NRBC cell count and critically ill patient´s outcome | 7 days
  The NRBC count will be obtained in first 7 days after admission. The NRBC count will be evaluated for the possibility correlation with the outcome (mortality and morbidity) of critically ill paediatric patients in PICU sepsis/septic shock?

CONTACTS AND LOCATIONS:
Overall Officials: Petr Dominik, MD., Principal Investigator — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651
- [Background] De Blasi RA, Cardelli P, Costante A, Sandri M, Mercieri M, Arcioni R. Immature platelet fraction in predicting sepsis in critically ill patients. Intensive Care Med. 2013 Apr;39(4):636-43. doi: 10.1007/s00134-012-2725-7. Epub 2012 Oct 24. PMID 23093245
- [Background] Nierhaus A, Klatte S, Linssen J, Eismann NM, Wichmann D, Hedke J, Braune SA, Kluge S. Revisiting the white blood cell count: immature granulocytes count as a diagnostic marker to discriminate between SIRS and sepsis--a prospective, observational study. BMC Immunol. 2013 Feb 12;14:8. doi: 10.1186/1471-2172-14-8. PMID 23398965
- [Background] Liu Y, Hou JH, Li Q, Chen KJ, Wang SN, Wang JM. Biomarkers for diagnosis of sepsis in patients with systemic inflammatory response syndrome: a systematic review and meta-analysis. Springerplus. 2016 Dec 12;5(1):2091. doi: 10.1186/s40064-016-3591-5. eCollection 2016. PMID 28028489
- [Background] Enz Hubert RM, Rodrigues MV, Andreguetto BD, Santos TM, de Fatima Pereira Gilberti M, de Castro V, Annichino-Bizzacchi JM, Dragosavac D, Carvalho-Filho MA, De Paula EV. Association of the immature platelet fraction with sepsis diagnosis and severity. Sci Rep. 2015 Jan 26;5:8019. doi: 10.1038/srep08019. PMID 25620275
- [Background] Schaer C, Schmugge M, Frey B. Prognostic value of nucleated red blood cells in critically ill children. Swiss Med Wkly. 2014 Mar 28;144:w13944. doi: 10.4414/smw.2014.13944. eCollection 2014. PMID 24706413
- [Background] Straney L, Clements A, Parslow RC, Pearson G, Shann F, Alexander J, Slater A; ANZICS Paediatric Study Group and the Paediatric Intensive Care Audit Network. Paediatric index of mortality 3: an updated model for predicting mortality in pediatric intensive care*. Pediatr Crit Care Med. 2013 Sep;14(7):673-81. doi: 10.1097/PCC.0b013e31829760cf. PMID 23863821
- [Background] Leteurtre S, Duhamel A, Salleron J, Grandbastien B, Lacroix J, Leclerc F; Groupe Francophone de Reanimation et d'Urgences Pediatriques (GFRUP). PELOD-2: an update of the PEdiatric logistic organ dysfunction score. Crit Care Med. 2013 Jul;41(7):1761-73. doi: 10.1097/CCM.0b013e31828a2bbd. PMID 23685639